CLINICAL TRIAL: NCT00993044
Title: A Phase I Study of Vincristine, Escalating Doses of Irinotecan, Temozolomide and Bevacizumab (Vit-b) in Pediatric and Adolescent Patients With Recurrent or Refractory Solid Tumors of Non-hematopoietic Origin
Brief Title: A Study of Vincristine, Escalating Doses of Irinotecan, Temozolomide and Bevacizumab (Vit-b) in Pediatric and Adolescent Patients With Recurrent or Refractory Solid Tumors of Non-hematopoietic Origin
Acronym: VIT-B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Leo Mascarenhas, Medical Staff/USC Faculty CWR, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-09-00214
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Refractory Solid Tumors in Children
MeSH Terms: interventions — Irinotecan; Vincristine; Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Irinotecan; Drug: Vincristine; Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Drug: Irinotecan — Dose Level 1 Irinotecan 30 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 1.5* Irinotecan 40 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 2 Irinotecan 50 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level -1 Irinotecan 20 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  * Dose escalation will proceed from dose level 1 to dose level 2 and de-escalate to dose level 1.5 if DLT is observed on dose level 2
Drug: Vincristine — Dose Level 1 Irinotecan 30 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 1.5* Irinotecan 40 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 2 Irinotecan 50 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level -1 Irinotecan 20 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  * Dose escalation will proceed from dose level 1 to dose level 2 and de-escalate to dose level 1.5 if DLT is observed on dose level 2
Drug: Temozolomide — Dose Level 1 Irinotecan 30 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 1.5* Irinotecan 40 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 2 Irinotecan 50 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level -1 Irinotecan 20 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  * Dose escalation will proceed from dose level 1 to dose level 2 and de-escalate to dose level 1.5 if DLT is observed on dose level 2
Drug: Bevacizumab — Dose Level 1 Irinotecan 30 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 1.5* Irinotecan 40 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 2 Irinotecan 50 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level -1 Irinotecan 20 mg/m2/day IV on day 1,2,3,4 and 5 Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  * Dose escalation will proceed from dose level 1 to dose level 2 and de-escalate to dose level 1.5 if DLT is observed on dose level 2

SUMMARY:
This phase I study is designed to determine the maximum tolerated dose of Irinotecan given intravenous for 5 days every 3 weeks in combination with fixed doses of Vincristine, Temozolomide and Bevacizumab (VIT-B) in patients with refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be > 12 months and < 21 years of age at the time of study entry.
* Weight: Patient must be more than or equal to 10 Kilograms.

Histological Diagnosis:

* Patients must have had histological verification of the malignancy at some time prior to study entry.
* All solid tumors are eligible with the exclusion of lymphomas. For patients with neuroblastoma, diagnosis based on elevated catecholamines in the urine and tumor cells on bone marrow aspirates/biopsies is acceptable.
* For patients with germ cell tumors, diagnosis based on elevated tumor markers (serum alpha fetoprotein and/or serum beta human chorionic gonadotropin) and radiographic evidence of disease is acceptable.

Disease Status:

* Disease must have failed standard therapy (therapies) or be a disease for which no standard therapy exists.
* Patient with stable disease on other therapies are not eligible.

Performance Level:

* Karnofsky > 50% for patients >16 years of age and Lansky > 50 for children < 16 years of age (Appendix I).
* Life Expectancy: Must be > 8 weeks.

Exclusion Criteria:

* Patients who have received bevacizumab and/or Irinotecan previously are ineligible. Non brain tumor patients who have previously received Temozolomide are ineligible.
* Pregnancy or Breast-Feeding: Pregnant patients are ineligible for this study due to the known teratogenic effects of the cytotoxic agents. Pregnancy tests must be obtained in females of childbearing potential prior to enrollment.
* Lactating women must agree not to breast-feed.
* Males or females of reproductive age may not participate unless they have agreed to use an effective contraceptive method.
* Patients Who Have an Uncontrolled Infection will not be eligible for enrollment until all infections are under control.
* Clinically Significant Unrelated Systemic Illness: Patients with serious infections or significant pulmonary, hepatic, renal, or other end-organ dysfunction which in the judgment of the Principal or Co-Investigators would compromise the patient's ability to tolerate prescribed chemotherapy or are likely to interfere with the study procedures or results will not be eligible.

Ages: 12 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajkumar Venkatramani, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Venkatramani R, Malogolowkin M, Davidson TB, May W, Sposto R, Mascarenhas L. A phase I study of vincristine, irinotecan, temozolomide and bevacizumab (vitb) in pediatric patients with relapsed solid tumors. PLoS One. 2013 Jul 22;8(7):e68416. doi: 10.1371/journal.pone.0068416. Print 2013. PMID 23894304

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: combination of Irinotecan, vincristine, temozolomide and bevacizumab: Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 1 Irinotecan 30 mg/m2/day IV on day 1,2,3,4 and 5
  Dose Level 1.5* Irinotecan 40 mg/m2/day IV on day 1,2,3,4 and 5
  Dose Level 2 Irinotecan 50 mg/m2/day IV on day 1,2,3,4 and 5
  Dose Level -1 Irinotecan 20 mg/m2/day IV on day 1,2,3,4 and 5
  * Dose escalation will proceed from dose level 1 to dose level 2 and de-escalate to dose level 1.5 if DLT is observed
Period: Irinotecan 30 mg
Arm/Group | Single Arm
Started | 6
Completed | 6
Not Completed | 0
Period: Irinotecan 50 mg
Arm/Group | Single Arm
Started | 7
Completed | 6
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dose Level 1, 2
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: Years] | 11 [3.9 to 19.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: Number of participants with dose limiting toxicity events
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 12
participants | 2

ADVERSE EVENTS:
Groups:
- Dose Level 1: combination of Irinotecan, vincristine, temozolomide and bevacizumab: Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 1 Irinotecan 30 mg/m2/day IV on day 1,2,3,4 and 5
- Dose Level 2: combination of Irinotecan, vincristine, temozolomide and bevacizumab: Vincristine 1.5mg/m2 (2mg max dose) IV on day 1,8 Temozolomide 100 mg/m2 PO on day 1,2,3,4 and 5 Bevacizumab 15mg/kg IV on day 1
  Dose Level 2 Irinotecan 50 mg/m2/day IV on day 1,2,3,4 and 5
Arm/Group | Dose Level 1 | Dose Level 2
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=6)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 — The first patient enrolled on dose level 1 had Noonan syndrome and recurrent synovial sarcoma.
colitis (Gastrointestinal disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=6)
Anemia (Blood and lymphatic system disorders) | 6 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No